CLINICAL TRIAL: NCT06066957
Title: Open Label Trial of Tolerability and Efficacy of Oral Letermovir for CMV Prophylaxis Among Heart and Lung Transplant Recipients
Brief Title: Open Label Trial of Oral Letermovir for CMV Prophylaxis in Thoracic Transplant Recipients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 853851
Record Dates: First submitted 2023-09-13; First posted 2023-10-04 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Cytomegalovirus Infections; Transplant-Related Disorder
Keywords: CMV; Thoracic Transplant
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — letermovir

STUDY DESIGN:
Intervention Model Description: This study is a prospective cohort design. Subjects exposed to letermovir for CMV prophylaxis following heart or lung transplantation will be compared with those who received standard valganciclovir prophylaxis in the two years before the study began (referred to as the "pre-intervention" period). The goal is to evaluate the efficacy and tolerability of letermovir.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Letermovir (Experimental): Will include those participants who receive letermovir for CMV prophylaxis as provided through the clinical trial. The "exposed" group will be ascertained prospectively over a one-year period (the "post-intervention" period).
  Interventions: Drug: Letermovir 480 MG [Prevymis]

INTERVENTIONS:
Drug: Letermovir 480 MG [Prevymis] — Letermovir for CMV prophylaxis in thoracic organ transplant recipients.
  Letermovir will be administered by oral administration, as per study protocol. The intended duration of therapy will be up to 365 days, depending on organ transplanted and donor and recipient CMV status. However, treatment may discontinued as discussed in Section 7.
  Letermovir is dosed at 480mg daily for patients with CrCl >10. Dose adjustment, as per package insert, is recommended in setting of co-administration of cyclosporine, with dose reduction of letermovir to 240mg daily. Missed doses of letermovir will not be made up.

SUMMARY:
Open label study to determine tolerability and efficacy of letermovir for CMV prophylaxis in heart and lung transplant recipients. The study hypotheses are:

1. Letermovir prophylaxis will be associated with similar rates of CMV infection as valganciclovir among heart and lung transplant recipients
2. Letermovir will be better tolerated than valganciclovir for CMV prophylaxis in heart and lung transplant recipients, with a higher proportion of days of completed therapy with correct dosing during the planned prophylaxis period
3. Letermovir will have a lower rate of neutropenia than valganciclovir when used for CMV prophylaxis in heart and lung transplant recipients
4. Incorrect renal dosing will occur less frequently with letermovir than with valganciclovir when used for CMV prophylaxis in heart and lung transplant recipients

DETAILED DESCRIPTION:
This study is a prospective cohort design. Subjects exposed to letermovir for CMV prophylaxis following heart or lung transplantation will be compared with those who received standard valganciclovir prophylaxis in the two years before the study began (referred to as the "pre-intervention" period). The goal is to evaluate the efficacy and tolerability of letermovir.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Age is >=18 years on the day of transplantation.
2. Heart or Lung transplant recipient.
3. Donor and/or Recipient CMV seropositive (defined by positive IgG) within 1 year prior to transplantation.
4. Able to start oral CMV prophylaxis within 14 days (heart graft recipients) or 28 days (lung graft recipients) of transplantation.
5. Males at birth agree to use contraception during the treatment period, and for at least 90 days after the last dose of study treatment, and refrain from donating sperm during this period.
6. Female at birth is not pregnant or breastfeeding. If of childbearing potential, agrees to follow the contraception guidance during the treatment period and for at least 90 days after the last dose of study treatment.
7. A male or female subject who is of reproductive potential agrees to true abstinence or to use (or have their partner use) 1 acceptable method of birth control starting from the time of consent through 90 days after the last dose of study therapy. True abstinence is defined as abstinence in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., abstinence only on certain calendar days, abstinence only during ovulation period, use of symptothermal method, use of post-ovulation methods) and withdrawal are not acceptable methods of contraception. Acceptable methods of birth control are: intrauterine device (IUD), diaphragm with spermicide, contraceptive sponge, condom, and vasectomy OR use of appropriate double barrier contraception as per local regulations or guidelines. Hormonal contraceptives (e.g., birth control pills, transdermal patch, or injectables) are unacceptable methods of birth control for use in this study because it is not known whether these methods are affected by co- administration of letermovir.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Any prior solid organ transplant.
2. Dual organ transplantation.
3. Prior treated CMV infection.
4. Unknown CMV serostatus of the donor or recipient.
5. Suspected or known hypersensitivity to active or inactive ingredients of letermovir formulations and/or acyclovir formulations.
6. CrCl <10 mL/minute, using Cockcroft-Gault equation, or renal replacement therapy at the time of enrollment.
7. Child-Pugh Class C severe hepatic insufficiency at enrollment.
8. Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 x the upper limit of normal (ULN) or serum total bilirubin > 2.5 x ULN. Note: Subjects who meet this exclusion criterion may, at the discretion of the investigator, have one repeat set of relevant labs done. If the repeat value does not meet this criterion, they may continue in the enrollment process.
9. Both moderate hepatic insufficiency AND moderate renal insufficiency. Note: Moderate hepatic insufficiency is defined as Child Pugh Class B; moderate renal insufficiency is defined as a creatinine clearance less than 50 mL/min, as calculated by the Cockcroft-Gault equation.
10. Neutropenia, defined as absolute neutrophil count <1,500/microliter, at the time of enrollment.
11. Severe thrombocytopenia, defined as platelets <50,000/microliter, at the time of enrollment.
12. Any uncontrolled infection on the day of enrollment.
13. Documented positive results for human immunodeficiency virus antibody (HIV-Ab) test at any time prior to enrollment, or hepatitis B surface antigen (HBsAg) within 90 days prior to enrollment.
14. Documented positive result for hepatitis C virus antibody (HCV-Ab) and with detectable HCV ribonucleic acid (RNA) within 90 days prior to enrollment with need for treatment with direct acting antiviral other than the following: glecaprevir/pibrentasvir, sofosbuvir/velpatasvir, or elbasvir/grazoprevir.
15. Pregnant or expecting to conceive, is breastfeeding, or plans to breastfeed from the time of consent through at least 90 days following cessation of study therapy.
16. Expecting to donate eggs or sperm starting from the time of consent through at least 90 days following cessation of study therapy.
17. Received within 30 days prior to enrollment or plans to receive during the study any of the following anti-CMV IgG antibody treatment or anti-CMV drug therapy including the following: Cidofovir, CMV hyper-immune globulin, any investigational CMV antiviral agent/biologic therapy.
18. Heart transplant recipients received >14 days of IV ganciclovir or oral valganciclovir prior to initiation of study drug or plans to receive during the study any of the following anti-CMV drug therapy: ganciclovir, valganciclovir, foscarnet. Lung transplant recipients received >28 days of IV ganciclovir or oral valganciclovir prior to initiation of study drug or plans to receive during the study any of the following anti-CMV drug therapy: ganciclovir, valganciclovir, foscarnet.
19. Currently participating or has participated in a study with an unapproved investigational compound within 28 days, or 5× half-life of the investigational compound whichever is longer, of initial dosing on this study.
20. Previously participated in this study or any other study involving letermovir.
21. Previously participated or is currently participating in any study involving administration of a CMV vaccine or another CMV investigational agent or is planning to participate in a study of a CMV vaccine or another CMV investigational agent during the course of this study.
22. For unexposed subjects, any letermovir exposure.
23. Are unable to take medications orally by day 14 post heart transplant or by day 28 post lung transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
CMV viral load | Prophylaxis period plus 180 days
  The primary outcome will be CMV infection (CMV viremia with CMV viral load >1,000, CMV syndrome, or tissue invasive CMV disease) during the planned prophylaxis period and the following 180 days
Proportion of days during which appropriately renally-dosed prophylaxis | 90 to 365 days post intervention
  The primary outcome will be the proportion of days during which appropriately-dosed prophylaxis was received during the planned treatment course.

SECONDARY OUTCOMES:
Biopsy-proven acute cellular rejection | Prophylaxis period plus 180 days
  The proportion of subjects who develop biopsy-proven acute cellular rejection
Proportion of subjects who develop CMV resistance | Prophylaxis period plus 180 days
  CMV resistance will be determined by the presence of a clinically significant mutation on genomic sequencing
Proportion of subjects who develop neutropenia | 90 to 365 days of prophylaxis period
  Proportion of subjects who develop Neutropenia (absolute neutrophil count (ANC) less than 1,500/microliter)
Proportion of subjects who develop severe thrombocytopenia (platelet count less than 50,000/microliter) | 90 to 365 days of prophylaxis period
  Proportion of subjects who develop severe thrombocytopenia (platelet count less than 50,000/microliter)
Proportion of subjects with Unplanned discontinuation of MMF or azathioprine | 90 to 365 days of prophylaxis period
  Proportion of subjects with Unplanned discontinuation of MMF or azathioprine
Number subjects with Incorrect renal dosing at any point during the planned prophylaxis period (measured as a binary variable, where the outcome is met if the recipient receives any days of incorrect dosing per their GFR). | 90 to 365 days of prophylaxis period
  Number subjects with Incorrect renal dosing at any point during the planned prophylaxis period (measured as a binary variable, where the outcome is met if the recipient receives any days of incorrect dosing per their GFR).

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Medicine at the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided